CLINICAL TRIAL: NCT05570487
Title: Increasing the Number of Resected Lymph Nodes Improves Overall Survival of Patients With Esophageal Squamous Cell Carcinoma With Positive Lymph Nodes: a Retrospective Analysis of 1656 Cases at a Single Cancer Center
Brief Title: RESECTED LYMPH NODES AND SURVIVAL OF PATIENTS WITH ESOPHAGEAL SQUAMOUS CELL CARCINOMA: AN OBSERVATIONAL STUDY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SichuanCHRIA
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: the Records of Esophageal Cancer
Keywords: esophageal cancer; lympha nodes
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- N0A Group: patients with negative lymph nodes and resected lymph nodes less than 15
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions
- N0B Group: patients with negative lymph nodes and resected lymph nodes no less than 15
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions
- N+A Group: patients with positive lymph nodes and resected lymph nodes less than 15
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions
- N+B Group: patients with positive lymph nodes and resected lymph nodes no less than 15
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions

INTERVENTIONS:
Diagnostic Test: Since the data were collected retrospectively, there were no interventions — Since the data were collected retrospectively, there were no interventions

SUMMARY:
To clarify the effect of the number of lymph node dissection and the number of stations on survival

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-85;
2. Histologically confirmed primary thoracic esophageal squamous cell carcinoma,
3. Staging PT1-4A, N0-3, M0 AJCC eighth edition;
4. Excluding lymph node dissection < 15,(meeting the guideline criteria)

Exclusion Criteria:

1. Patients with a history of previous thoracic and abdominal surgery that may affect lymphatic reflux
2. Patients with distant metastasis confirmed by imaging;
3. Patients with obvious surgical contraindications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer and need surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The number of lymph nodes | 2010.1.1-2017.12.30
  Surgical data were retrospectively collected

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share data, analytic methods, and study materials related to this article with other researchers. Provided that all of the above will not be used for commercial or profit purposes. Other researchers can contact the corresponding author of this article by email and indicate the required research materials and purpose. We will be glad to provide relevant materials for this study after approval and discussion.

REFERENCES:
- [Derived] Li K, Leng X, Peng L. Resected lymph nodes and survival of patients with esophageal squamous cell carcinoma in pT2 and pT3. Int J Surg. 2024 Mar 1;110(3):1879-1881. doi: 10.1097/JS9.0000000000001023. No abstract available. PMID 38116658
- [Derived] Li K, Leng X, He W, Du K, Li C, Liu K, Wang C, Liu G, Li Z, Jiang L, Li K, Zhou Q, Li J, Luo X, Nie X, Lu S, Li H, Fang Q, Xiao W, Han Y, Peng L. Resected lymph nodes and survival of patients with esophageal squamous cell carcinoma: an observational study. Int J Surg. 2023 Jul 1;109(7):2001-2009. doi: 10.1097/JS9.0000000000000436. PMID 37222685